CLINICAL TRIAL: NCT01373489
Title: Effectiveness of Technology-Assisted Case Management in Low Income Adults With Type 2 Diabetes
Brief Title: Technology-assisted Case Management in Adults With Type 2 Diabetes
Acronym: TACM-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00009204; Department of Defense (Other Grant/Funding Number: W81XWH-10-2-0057)
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes
Keywords: type 2 diabetes; nurse case management; telemedicine
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The usual care group received the current standards of care at the study clinics.
- Technology Assisted Case Management (Experimental): The TACM group used the FORA 2-in-1 Telehealth system for diabetes management intervention to link a case manager to patients with poorly controlled type 2 diabetes in real time.
  Interventions: Behavioral: Technology-Assisted Case Management

INTERVENTIONS:
Behavioral: Technology-Assisted Case Management — The TACM intervention uses the FORA 2-in-1 Telehealth System for diabetes to link a case manager to poorly controlled diabetics in real time. Patients will be assigned the FORA 2-in-1 Telehealth System and provided glucose test strips to allow testing at least once a day. They will be asked to perform glucose testing and blood pressure measurement using the FORA system once daily. They will be asked to upload the measurements daily as soon as possible after the test is performed. The nurse case manager will have access to a secure server to which the uploaded measurements are stored in real time. Medications are titrated under supervision of a primary care and endocrinology physicians
  Arms: Technology Assisted Case Management

SUMMARY:
The purpose of this study is to help low income patients achieve and maintain better self-management skills and improve blood sugar levels, using a 2-in-1 blood glucose and blood pressure monitoring system and nurse case management. Patients must be served at a Federally Qualified Health Center (FQHC) in coastal South Carolina.

DETAILED DESCRIPTION:
The long-term goal is to develop a practical and sustainable system of diabetes management that will help low income patients achieve and maintain goals within established treatment guidelines regardless of geographic location. This randomized clinical trial will employ the innovative FORA system, an inexpensive, off-the-shelf, state-of-the-art technology comprised of a 2-in-1 Blood Glucose and Blood Pressure monitor, coupled with nurse case management (TACM) to optimize diabetes care for low income, rural adults with type 2 diabetes (T2DM). The target population will be low income patients served in Federally Qualified Health Care Centers (FQHCs) with poorly controlled T2DM residing in coastal South Carolina. Two hundred patients will be randomly assigned to two groups of 100 patients each; Group A (Usual Care) and Group B (Technology-assisted Case Management, TACM). Each patient will be followed for 6 months, with study visits at baseline, 3, and 6 months. The primary outcome will be Hemoglobin A1c (HbA1c) at 6 months post-randomization while the secondary outcomes will be blood pressure control and quality of life (qol) at 6 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and receiving care within the Franklin C. Fetter Family Health Center
* Clinical diagnosis of T2DM and HbA1c ≥8% at the screening visit
* Subject must be willing to use the FORA 2-in-1 system
* Subject must have a working land-line for the duration of the study in order to be able to upload the readings from the FORA 2-in-1 machine
* Subjects must be able to communicate in English

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Participation in other diabetes clinical trials
* Alcohol or drug abuse/dependency using a screening questionnaire
* Active psychosis or acute mental disorder
* Life expectancy <6 months
* Pregnant and/or lactating females

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Franklin C. Fetter Family Health Center, Inc., Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egede LE, Strom JL, Fernandes J, Knapp RG, Rojugbokan A. Effectiveness of technology-assisted case management in low income adults with type 2 diabetes (TACM-DM): study protocol for a randomized controlled trial. Trials. 2011 Oct 20;12:231. doi: 10.1186/1745-6215-12-231. PMID 22014122
- [Result] Egede LE, Williams JS, Voronca DC, Knapp RG, Fernandes JK. Randomized Controlled Trial of Technology-Assisted Case Management in Low Income Adults with Type 2 Diabetes. Diabetes Technol Ther. 2017 Aug;19(8):476-482. doi: 10.1089/dia.2017.0006. Epub 2017 Jun 5. PMID 28581821
- See also: Protocol Paper — https://pubmed.ncbi.nlm.nih.gov/22014122/
- See also: Primary Outcomes Paper — https://pubmed.ncbi.nlm.nih.gov/28581821/

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Typical office-based practice. In this setting the patient is custodian of his/her own care. Between scheduled visits, the patient is responsible for complying with prescribed treatment including medications, diet and exercise regimen, blood glucose monitoring, and follow up visits. Contact between scheduled visits is patient-initiated and occurs when the patient perceives a problem with the treatment plan. For patients with poorly controlled T2DM, which is often asymptomatic prior to the onset of serious complications, this is a particularly ineffective strategy.
- Technology-assisted Case Management (TACM): This model capitalizes on information technology like the FORA system to link a case manager to poorly controlled diabetics in real time. Clearly a model that is applicable only to patients in need of intensive intervention, the advantages includes accurate data transfer to a medical decision maker and positive reinforcement/feedback to the patient via the FORA system to enhance adherence. If the case manager has physician-supervised prescriptive authority, then medication adjustments can be made daily or weekly, if needed, to achieve and maintain control. More frequent interventions, combined with improved compliance with medications and testing frequency, the strategies that are known to work, are enabled by this approach.
  Technology-Assisted Case Management (TACM with the FORA 2-in-1 Telehealth System): The TACM intervention uses the FORA 2-in-1 Telehealth System for diabetes to link a case manager to poorly controlled diabetics in real time.
Period: Overall Study
Arm/Group | Usual Care | Technology-assisted Case Management (TACM)
Started | 59 | 54
Completed | 44 | 41
Not Completed | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Technology-assisted Case Management (TACM) | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 54 | 113
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 92
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 39 | 85
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 6 Months Post Randomization
Description: Hemoglobin A1c (HbA1c) was measured at 6 months post randomization
Time Frame: 6 months post randomization
Population: Final analysis used baseline A1c analysis of covariance for differences in levels of A1c at 6 months between the treatment groups with baseline A1c as covariate.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Usual Care | Technology-assisted Case Management (TACM)
Number analyzed (Participants) | 59 | 54
percentage of glycosylated hemoglobin | 10.0 (2.7) | 9.0 (1.9)
Statistical Analysis 1: Comparison: Usual Care vs Technology-assisted Case Management (TACM); Test type: Superiority; p < 0.05, ANCOVA; Mean Difference (Final Values) = 10

ADVERSE EVENTS:
Time Frame: 6month
Groups:
- Technology-assisted Case Management (TACM): This model capitalizes on information technology like the FORA system to link a case manager to poorly controlled diabetics in real time. Clearly a model that is applicable only to patients in need of intensive intervention, the advantages includes accurate data transfer to a medical decision maker and positive reinforcement/feedback to the patient via the FORA system to enhance adherence. If the case manager has physician-supervised prescriptive authority, then medication adjustments can be made daily or weekly, if needed, to achieve and maintain control. More frequent interventions, combined with improved compliance with medications and testing frequency, the strategies that are known to work, are enabled by this approach.
  Technology-Assisted Case Management (TACM with the FORA 2-in-1 Telehealth System): The TACM intervention uses the FORA 2-in-1 Telehealth System for diabetes to link a case manager to poorly controlled diabetics in real time. Patients assigned the FORA 2-
Arm/Group | Usual Care | Technology-assisted Case Management (TACM)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/54
Other Adverse Events (participants affected / at risk) | 0/59 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No